CLINICAL TRIAL: NCT04688775
Title: Interventional, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Delayed-Start Study to Evaluate the Efficacy and Safety of Eptinezumab in Patients With Episodic Cluster Headache
Brief Title: Eptinezumab in Participants With Episodic Cluster Headache
Acronym: ALLEVIATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19386A
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Cluster Headache, Episodic
MeSH Terms: conditions — Cluster Headache | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1: Eptinezumab Then Placebo (Experimental): Eptinezumab in the Placebo-controlled Period, followed by administration of placebo in the Active Treatment Period
  Interventions: Drug: Eptinezumab; Drug: Placebo
- Sequence 2: Placebo Then Eptinezumab (Experimental): Placebo in the Placebo-controlled Period, followed by administration of eptinezumab in the Active Treatment Period
  Interventions: Drug: Eptinezumab; Drug: Placebo

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab - concentrate for solution for infusion, intravenously
Drug: Placebo — Placebo - 100 milliliters (mL) of 0.9% normal saline, intravenously

SUMMARY:
The purpose of this study is to evaluate the efficacy of eptinezumab in participants with episodic Cluster Headache (eCH)

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned to receive treatment, in a blinded manner, two infusions of either eptinezumab or placebo in a cross-over manner during the Placebo-controlled Period and Active Treatment Period of the study.

The total duration of the study after randomization is 24 weeks, including a safety follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has episodic cluster headache, as defined by International Headache Society (IHS) International Classification of Headache Disorders 3rd Edition (ICHD-3) classification, with an adequately documented record or reliable history of eCH of at least 12 months prior to Screening Visit 1.
* The participant has a prior history of cluster period(s) lasting 6 weeks or longer, when untreated.
* The participant is able to distinguish cluster headache attacks from other headaches (that is; tension-type headaches, migraine).
* The participant is, at Screening Visit 2, in cluster headache bout, characterized by the presence of at least one typical cluster headache attack, that started not later than 1 week prior to Screening Visit 2.
* The participant has a medical history of first symptoms of cluster headache from ≤60 years of age.

Exclusion Criteria

* The participant has experienced failure on a previous treatment targeting the calcitonin gene-related peptide (CGRP) pathway (anti-CGRP monoclonal antibodies [mAbs] and gepants).
* The participant has confounding and clinically significant pain syndromes (for example, fibromyalgia, complex regional pain syndrome).
* The participant has a history or diagnosis of hypnic headache, hemicrania continua, new daily persistent headache, chronic migraine or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), recurrent painful ophthalmoplegic neuropathy, migraine with brainstem aura and migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration).
* Participants with a lifetime history of psychosis, bipolar mania, or dementia are excluded. Participants with other psychiatric conditions whose symptoms are not controlled or who have not been adequately treated for a minimum of 6 months prior to Screening Visit 2 are also excluded.
* The participant is, at Screening Visit 2, at significant risk of suicide.
* The participant has a history of clinically significant cardiovascular disease, including uncontrolled hypertension, ischaemia or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (120):
- United States (24):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic in Arizona - Phoenix Campus, Phoenix, Arizona
  - Keck School of Medicine of USC, Los Angeles, California
  - Clinical Research Institute, Los Angeles, California
  - Stanford Neurosciences Health Center, Palo Alto, California
  - Neurology Colorado - Denver Advanced Neurological Evaluation and Treatment Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Accel Research Sites - Tampa, Tampa, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Headache Center Mississippi, Ridgeland, Mississippi
  - Clinvest Research, Springfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - New York University School of Medicine, New York, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Cleveland Clinic - Neurological Institute, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital - Center City Campus, Philadelphia, Pennsylvania
  - Mischer Neuroscience Institute, Houston, Texas
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - Centre Hospitalier Chretien - Clinique MontLégia, Liège
- Czechia (4):
  - Mestska Nemocnice Ostrava, Ostrava, Moravian-Silesian
  - Fakultní Thomayerova nemocnice, Prague, Prague
  - FORBELI s.r.o. Neurologicka Ambulance, Prague, Prague
  - Institut Neuropsychiatrické Péce, Prague, Prague
- Denmark (4):
  - Rigshospitalet Glostrup, Glostrup Municipality, Capital Region
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
  - Hospitalsenhed Midt og Regionshospitalet Viborg, Viborg, Central Jutland
  - Sydvestjysk Sygehus - Esbjerg, Esbjerg
- Estonia (3):
  - Confido Meditsiinikeskus, Tallinn, Harju
  - Ida-Viru Keskhaigla, Kohtla-Järve, Ida-Virumaa
  - Tartu Ülikooli Kliinikum, Tartu, Tartu
- Finland (4):
  - Tampereen Yliopistollinen Sairaala (TAYS), Tampere, Länsi-Suomen Lääni
  - Terveystalo Ruoholahti, Helsinki, Southern Finland
  - Terveystalo Turku Pulssi, Turku, Western Finland
  - Terveystalo Tampere, Tampere
- France (8):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Centre Hospitalier Annecy Genevois, Metz-Tessy, Auvergne-Rhône-Alpes
  - Hôpital Cimiez, Nice, Côte-d'Or
  - Hôpital Roger Salengro, Lille, Nord
  - Hôpital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Priest-en-Jarez, Rhône
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital Lariboisière, Paris, Île-de-France Region
- Georgia (5):
  - Pineo Medical Ecosystem, Tbilisi
  - Archangel Saint Michael Multiprofile Clinical Hospital, Tbilisi
  - Aversi Clinic - Central Branch, Tbilisi
  - Simon Khechinashvili University Hospital, Tbilisi
  - Consilium Medulla Multiprofile Clinic, Tbilisi
- Germany (10):
  - Universität Heidelberg, Heidelberg, Baden-Wurttemberg
  - LMU Klinikum - Campus Grosshadern, München, Bavaria
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Western-Pommerania
  - Neurologische Praxis Dr. Stude, Bochum, North Rhine-Westphalia
  - Praxis für Neurologie, Psychosomatik, Nervenheilkunde, Psychotherapie und Spezielle Schmerztherapie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Schmerzklinik Kiel, Kiel, Schleswig-Holstein
  - Charité Campus Mitte, Berlin
- Greece (6):
  - 401 General Military Hospital of Athens, Athens, Attica
  - Eginition University - General Hospital of Athens, Athens, Attica
  - Mediterraneo Hospital, Glyfada, Attica
  - University General Hospital of Larissa, Larissa, Thessaly
  - General Hospital of Patras Agios Andreas, Pátrai, West Greece
  - Euromedica General Clinic - Thessaloniki, Thessaloniki
- Italy (10):
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - San Raffaele Pisana, Rome, Roma
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari, Bari
  - IRCCS Istituto Delle Scienze Neurologiche di Bologna, Bologna
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Fondazione Istituto Neurologico Car..., Milan
  - Azienda Ospedaliero - Universitaria di Modena, Modena
  - Azienda Ospedaliera Universitaria - Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Fondazione Mondino - Istituto Neurologico Nazionale a Carattere Scientifico IRCCS, Pavia
  - Universita Campus Bio-Medico di Roma, Rome
  - Ospedale Molinette - Clinica Neurologica II - Centro Cefalee, Turin
- Japan (3):
  - Sendai Headache And Neurology Clinic, Sendai, Miyagi
  - Saitama Neuropsychiatric Institute, Saitama-shi, Saitama
  - Japanese Red Cross Shizuoka Hospital, Shizuoka, Shizuoka
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Zuyderland Medisch Centrum Sittard-Geleen, Geleen, Limburg
  - Brain Research Center - Amsterdam, Amsterdam, North Holland
- Norway (2):
  - Oslo Hodepinesenter, Oslo
  - St. Olavs Hospital - Universitetssykehuset I Trondheim, Trondheim
- Portugal (4):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora, Lisbon District
  - Centro Hospitalar Universitario Lisboa Norte, E.P.E - Hospital De Santa Maria, Lisbon, Lisbon District
  - Hospital Garcia de Orta, Almada, Setúbal District
  - Hospital da Luz, Lisbon
- Russia (6):
  - City Hospital No. 33 of the Leninsky District of the city of Nizhny Novgorod, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Perm State Medical University named after E. A. Wagner of the Ministry of Healthcare of the Russi..., Perm, Permsky
  - Kazan State Medical University, Kazan', Tartarstan
  - First Moscow State Medical University named after I.M. Sechenov, Moscow
  - University Headache Clinic, Moscow
  - LLC Scientific and Practical Medical Center Innovation and Health, Novosibirsk
- Spain (11):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen Macarena, Castilleja de la Cuesta, Sevilla
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Sweden (5):
  - Hallands sjukhus Halmstad, Halmstad, Halland County
  - Skåneuro Privatmottagning, Lund, Skåne County
  - Karolinska Universitetssjukhuset Huddinge, Huddinge, Stockholm County
  - Danderyds Sjukhus, Stockholm, Stockholm County
  - Centralsjukhuset Karlstad, Karlstad, Värmland County
- United Kingdom (5):
  - Hull University Teaching Hospitals NHS Trust, Hull, England
  - The Walton Centre NHS Foundation Trust, Liverpool, England
  - King's College Hospital NHS Foundation Trust, London, England
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - Northern Care Alliance NHS Foundation Trust, Salford, England

REFERENCES:
- [Derived] Jensen RH, Tassorelli C, Tepper SJ, Charles A, Goadsby PJ, Snoer AH, Sperling B, Krog Josiassen M, Borgen Linander C, Ettrup A, Boneva N. Efficacy and Safety of Eptinezumab in Episodic Cluster Headache: A Randomized Clinical Trial. JAMA Neurol. 2025 Jul 1;82(7):706-714. doi: 10.1001/jamaneurol.2025.1317. PMID 40388178

RESULTS

PARTICIPANT FLOW:
Groups:
- Eptinezumab: Participants received a single intravenous (IV) infusion of eptinezumab 400 milligrams (mg) in 100 milliliters (mL) 0.9% saline solution.
- Placebo: Participants received a single IV infusion of 0.9% saline solution as matching placebo for eptinezumab.
- Delayed Start Period: Placebo to Eptinezumab: Participants who received eptinezumab in the placebo-controlled period received a single IV infusion of 0.9% saline solution as matching placebo for eptinezumab.
- Delayed Start Period: Eptinezumab to Placebo: Participants who received placebo in the placebo-controlled period received a single IV infusion of eptinezumab 400mg in 100 mL 0.9% saline solution.
Period: Placebo-controlled Period
Arm/Group | Eptinezumab | Placebo | Delayed Start Period: Placebo to Eptinezumab | Delayed Start Period: Eptinezumab to Placebo
Started | 113 | 118 | 0 | 0
Received at Least 1 Dose of Study Drug | 112 | 117 | 0 | 0
Completed | 108 | 107 | 0 | 0
Not Completed | 5 | 11 | 0 | 0
Not completed — Randomized, not treated | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 6 | 0 | 0
Not completed — Other reasons | 0 | 1 | 0 | 0
Period: Delayed Start Period
Arm/Group | Eptinezumab | Placebo | Delayed Start Period: Placebo to Eptinezumab | Delayed Start Period: Eptinezumab to Placebo
Started | 0 | 0 | 107 | 108
Received at Least 1 Dose of Study Drug | 0 | 0 | 107 | 108
Completed | 0 | 0 | 101 | 100
Not Completed | 0 | 0 | 6 | 8
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — other reasons | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The all-participants-randomized-set (APRS) included all randomized participants. The all-participants-treated set (APTS) included all randomized participants who received infusion with double-blind investigational medicinal product (IMP). Demographic characteristics were collected for the APTS and study-specific characteristics were collected for the APRS.
Groups:
- Eptinezumab: Participants received a single IV infusion of eptinezumab 400mg in 100 mL 0.9% saline solution.
- Total: Total of all reporting groups
Arm/Group | Eptinezumab | Placebo | Total
Number analyzed (Participants) | 113 | 118 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The APTS included all randomized participants in the who received infusion with double-blind IMP.
  years
    number analyzed (Participants) | 112 | 117 | 229
    (all) | 44.17 (11.099) | 43.94 (11.019) | 44.05 (11.035)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The APTS included all randomized participants who received infusion with double-blind investigational medicinal product (IMP).
  Participants
    number analyzed (Participants) | 112 | 117 | 229
    Female | 27 | 24 | 51
    Male | 85 | 93 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The APTS included all randomized participants in the who received infusion with double-blind IMP.
  Participants
    number analyzed (Participants) | 112 | 117 | 229
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 4 | 4 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 97 | 103 | 200
    Other | 1 | 2 | 3
    Unknown or Not Reported | 9 | 8 | 17
Number of Weekly Cluster Headache (CH) Attacks [Mean (Standard Deviation); unit: Number of Weekly Attacks] — Population: The APRS included all randomized participants.
  Number of Weekly Attacks | 15.2 (8.07) | 15.7 (8.28) | 15.4 (8.17)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Weekly Cluster Headache (CH) Attacks, Averaged Over Weeks 1-2
Description: The participant completed a CH eDiary, daily, and recorded for each day/week whether he/she had any CH attacks. For each CH attack, the start date and time was collected. The participant recorded further daily information regarding CH characteristics and intake of acute medication for CH. CH items were assessed with a yes/no response.
Time Frame: Baseline (Week 0), Weeks 1-2
Population: The APRS included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Number of Weekly Attacks
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 113 | 118
Number of Weekly Attacks | -4.0 (0.93) | -4.6 (0.89)
Statistical Analysis 1: Comparison: Eptinezumab vs Placebo; Change From Baseline in the Number of Weekly Attacks: Eptinezumab vs. Placebo; Test type: Superiority; p = 0.5048, Mixed Models Repeated Measures; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.3 to 2.6]

2. Secondary Outcome: Number of Participants With ≥50% Reduction From Baseline in Number of Weekly Attacks Over Weeks 1-2
Time Frame: Baseline (Week 0), Weeks 1-2
Population: The APRS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 113 | 118
Participants | 44 | 37

3. Secondary Outcome: Change From Baseline in the Number of Weekly Times an Abortive Medication Was Used, Averaged Over Weeks 1-2
Description: Abortive medications included the use of triptans or oxygen (O2).
Time Frame: Baseline (Week 0), Weeks 1-2
Population: The APRS included all randomized participants. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Abortive therapy use per week
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
Abortive therapy use per week | -2.54 (0.98) | -3.55 (0.93)

4. Secondary Outcome: Change From Baseline in the Number of Daily Attacks, Averaged Over Days 1-3
Time Frame: Baseline (Week 0), Days 1-3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Attacks per day
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 110 | 115
Attacks per day | -0.22 (0.16) | -0.35 (0.15)

5. Secondary Outcome: Change From Baseline in the Number of Days With <3 Attacks Per Day, Averaged Over Weeks 1-2
Time Frame: Baseline (Week 0), Weeks 1-2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
Days | 0.60 (0.20) | 0.82 (0.19)

6. Secondary Outcome: Time From First Infusion of IMP to Resolution of Cluster Headache Bout Within the First 4 Weeks
Description: Presented here is the result of the analysis of time from first infusion of IMP to resolution of cluster headache bout. The hazard ratio estimate is an estimate from the Cox model of time to resolution.
Time Frame: From first infusion (Baseline, Day 0) to 4 weeks
Population: The APRS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 112 | 117
days | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of events | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of events
Statistical Analysis 1: Comparison: Eptinezumab vs Placebo; Test type: Superiority; p = 0.0772, Regression, Cox; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.96 to 2.17]

7. Secondary Outcome: Change From Baseline in Number of Attacks Starting ≤24 Hours After the Start of the First Infusion of IMP
Time Frame: From first infusion in the placebo-controlled period (Baseline, Day 0) to 24-hours after the first infusion in the placebo-controlled period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Number of attacks
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 104 | 110
Number of attacks | 2.07 (0.18) | 1.96 (0.17)

8. Secondary Outcome: Change From Baseline in the Daily Mean Score on 5-Point Self-Rating Pain Severity Scale, Averaged Over Days 1-3
Description: The severity of pain was rated on an ordinal scale that ranged from 0 to 4 with higher scores indicating more headache pain (headache pain ratings: 0 = none/barely any pain; 1 = mild; 2 = moderate; 3 = severe; 4 = excruciating).
Time Frame: Baseline (Week 0), Days 1-3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 99 | 112
score on a scale | -0.30 (0.10) | -0.18 (0.09)

9. Secondary Outcome: Change From Baseline to Week 1 in the Number of Weekly Attacks
Time Frame: Baseline (Week 0), Week 1
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
Attacks per week | -2.62 (0.95) | -3.71 (0.90)

10. Secondary Outcome: Change From Baseline to Week 2 in the Number of Weekly Attacks
Time Frame: Baseline (Week 0), Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 106 | 110
Attacks per week | -5.44 (1.00) | -5.64 (0.96)

11. Secondary Outcome: Number of Participants With ≥50% Reduction From Baseline in Number of Weekly Attacks in Week 1
Time Frame: Baseline (Week 0), Week 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
Participants | 36 | 28

12. Secondary Outcome: Number of Participants With ≥30% Reduction From Baseline in Number of Weekly Attacks in Week 1
Time Frame: Baseline (Week 0), Week 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
Participants | 48 | 50

13. Secondary Outcome: Number of Participants With ≥30% Reduction From Baseline in Number of Weekly Attacks Over Weeks 1-2
Time Frame: Baseline (Week 0), Weeks 1-2
Population: The APRS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 113 | 118
Participants | 59 | 53

14. Secondary Outcome: Change From Baseline in Weekly Integrated Measure of Frequency and Intensity of Pain, Averaged Over Weeks 1-2
Description: The weekly integrated measure of frequency and intensity of pain calculates a singular numerical value for frequency and intensity of pain by adding the intensity rating (Worst pain on a 5-point Self-rating pain severity scale) for each attack during that week. The intensity of pain for each attack was rated on an ordinal scale that ranged from 0 to 4 with higher scores indicating more headache pain (0 = none/barely any pain; 1 = mild; 2 = moderate; 3 = severe; 4 = excruciating). The total weekly score could range from 0 (no attacks and/or no pain) to no specified upper limit, with lower scores representing better outcomes.
Time Frame: Baseline (Week 0), Weeks 1-2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
score on a scale | -13.39 (2.56) | -14.46 (2.43)

15. Secondary Outcome: Change From Baseline to Week 1 in Weekly Integrated Measure of Frequency and Intensity of Pain
Description: as for outcome 14
Time Frame: Baseline (Week 0), Week 1
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
score on a scale | -10.58 (2.55) | -11.96 (2.42)

16. Secondary Outcome: Change From Baseline to Week 2 in Weekly Integrated Measure of Frequency and Intensity of Pain
Description: as for outcome 14
Time Frame: Baseline (Week 0), Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 106 | 110
score on a scale | -16.20 (2.73) | -16.95 (2.61)

17. Secondary Outcome: Change From Baseline in the Number of Weekly Attacks, Averaged Over Weeks 1-4
Time Frame: Baseline (Week 0), Weeks 1-4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
Attacks per week | -5.95 (0.92) | -5.78 (0.88)

18. Secondary Outcome: Change From Baseline in Weekly Integrated Measure of Frequency and Intensity of Pain, Averaged Over Weeks 1-4
Description: The weekly integrated measure of frequency and intensity of pain score calculates a singular numerical value for frequency and intensity of pain by adding the intensity rating (Worst pain on a 5-point Self-rating pain severity scale) for each attack during that week. The intensity of pain for each attack was rated on an ordinal scale that ranged from 0 to 4 with higher scores indicating more headache pain (0 = none/barely any pain; 1 = mild; 2 = moderate; 3 = severe; 4 = excruciating). The total weekly score could range from 0 (no attacks and/or no pain) to no specified upper limit, with lower scores representing better outcomes.
Time Frame: Baseline (Week 0), Weeks 1-4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 109 | 116
score on a scale | -17.81 (2.50) | -16.81 (2.37)

19. Secondary Outcome: Change From Baseline in the Mean Score on 5-Point Self-Rating Pain Severity Scale (Average Per Attack Over a Week) for Weeks 1, 2, 3, and 4
Description: The severity of pain for each attack was rated on an ordinal scale that ranged from 0 to 4 with higher scores indicating more headache pain (headache pain ratings: 0 = none/barely any pain; 1 = mild; 2 = moderate; 3 = severe; 4 = excruciating).
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, and 4
Population: The APRS included all randomized participants. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure and "Number Analyzed" is the number of participants evaluable at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 101 | 116
score on a scale
  Week 1 | -0.33 (0.09) | -0.24 (0.08)
  Week 2: number analyzed (Participants) | 91 | 100
  Week 2 | -0.46 (0.10) | -0.35 (0.09)
  Week 3: number analyzed (Participants) | 80 | 97
  Week 3 | -0.56 (0.11) | -0.31 (0.10)
  Week 4: number analyzed (Participants) | 70 | 86
  Week 4 | -0.51 (0.11) | -0.42 (0.10)

20. Secondary Outcome: Change From Baseline in the Number of Weekly Attacks for Each of Weeks 3 and 4
Time Frame: Baseline (Week 0), Weeks 3-4
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 104 | 112
Attacks per week
  Week 3 | -7.35 (0.98) | -6.60 (0.94)
  Week 4: number analyzed (Participants) | 102 | 107
  Week 4 | -8.37 (1.11) | -7.15 (1.07)

21. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Weeks 1, 2, and 4
Description: The PGIC is a patient-reported measure of improvement in pain sensation and quality of life scored on a scale from 1 (very much improved) to 7 (very much worse). Lower scores indicate better health status.
Time Frame: Weeks 1, 2, and 4
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 104 | 106
score on a scale
  Week 1: number analyzed (Participants) | 102 | 96
  Week 1 | 3.19 (0.16) | 3.55 (0.15)
  Week 2: number analyzed (Participants) | 95 | 93
  Week 2 | 2.92 (0.17) | 3.44 (0.16)
  Week 4 | 2.85 (0.18) | 3.23 (0.17)

22. Secondary Outcome: Change From Baseline in Sleep Impact Scale (SIS) Domain Scores at Weeks 2 and 4
Description: The SIS is a patient-reported clinical outcome assessment used to assess quality of life resulting from sleep disturbance. The SIS questionnaire includes 35 items belonging to 7 domains to assess sleep impact on: daily activities; emotional well-being; emotional impact; energy/fatigue; social well-being; mental fatigue; and satisfaction with sleep. Each item, for 6 out of the 7 domains, is rated on a 5-point scale ranging from 1 (always or all of the time) to 5 (never or none of the time), whereas satisfaction with sleep is rated on a 5-point scale ranging from 1 (very satisfied) to 5 (very dissatisfied). Each domain yields a score ranging from 0 to 100, which is presented here. A higher score for Daily Activities, Emotional Well-being, Emotional Impact, Energy/Fatigue, Social Well-being, and Mental Fatigue indicates better quality of life. A lower score for Satisfaction with Sleep indicates a higher quality of life.
Time Frame: Baseline (Week 0), Weeks 2 and 4
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 100 | 102
score on a scale
  Daily Activities - Week 2: number analyzed (Participants) | 91 | 84
  Daily Activities - Week 2 | 16.83 (3.08) | 8.93 (3.06)
  Daily Activities - Week 4 | 24.82 (3.19) | 13.97 (3.08)
  Emotional Well-being - Week 2: number analyzed (Participants) | 91 | 84
  Emotional Well-being - Week 2 | 14.85 (2.84) | 6.04 (2.81)
  Emotional Well-being - Week 4 | 22.77 (3.07) | 12.22 (2.97)
  Energy/Fatigue - Week 2: number analyzed (Participants) | 91 | 84
  Energy/Fatigue - Week 2 | 18.16 (3.23) | 8.03 (3.19)
  Energy/Fatigue - Week 4 | 24.16 (3.47) | 14.68 (3.36)
  Mental Fatigue - Week 2: number analyzed (Participants) | 91 | 84
  Mental Fatigue - Week 2 | 9.04 (2.66) | 4.15 (2.64)
  Mental Fatigue - Week 4 | 15.15 (2.91) | 8.00 (2.81)
  Emotional Impact - Week 2: number analyzed (Participants) | 91 | 84
  Emotional Impact - Week 2 | 14.39 (3.02) | 6.00 (3.00)
  Emotional Impact - Week 4 | 23.09 (3.29) | 13.36 (3.18)
  Social Well-being - Week 2: number analyzed (Participants) | 91 | 84
  Social Well-being - Week 2 | 15.22 (3.37) | 6.92 (3.35)
  Social Well-being - Week 4 | 23.74 (3.46) | 13.91 (3.35)
  Satisfaction with Sleep - Week 2: number analyzed (Participants) | 91 | 84
  Satisfaction with Sleep - Week 2 | -11.41 (2.75) | -6.06 (2.73)
  Satisfaction with Sleep - Week 4 | -19.60 (2.88) | -9.63 (2.78)

23. Secondary Outcome: Change From Baseline in Euroqol 5-Dimension 5-Levels (EQ-5D-5L) Visual Analogue Scale (VAS) at Weeks 2 and 4
Description: The EQ-5D-5L VAS is a participant-reported assessment designed to measure the participant's well-being and ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline (Week 0), Weeks 2 and 4
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 76 | 80
score on a scale
  Week 2: number analyzed (Participants) | 70 | 63
  Week 2 | 8.21 (2.79) | 3.47 (2.86)
  Week 4 | 13.49 (2.80) | 5.73 (2.77)

24. Secondary Outcome: Health Care Resource Utilization (HCRU) Score: Number of Visits to a Family Doctor/General Practitioner
Description: Number of participants who visited a family doctor/general practitioner has been reported.
Time Frame: Week 4
Population: The APRS included all randomized participants. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 100 | 104
Participants
  0 visits | 85 | 85
  1 visit | 9 | 10
  2 visits | 1 | 6
  3 visits | 3 | 1
  5 visits | 1 | 1
  6 visits | 1 | 1

25. Secondary Outcome: HCRU Score: Number of Visits to a Specialist
Description: Number of participants who visited a specialist has been reported.
Time Frame: Week 4
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 100 | 104
Participants
  0 visits | 77 | 68
  1 visit | 11 | 18
  2 visits | 6 | 14
  3 visits | 4 | 2
  4 visits | 2 | 2

26. Secondary Outcome: HCRU Score: Number of Emergency Department Visits Due to Cluster Headache
Description: Number of participants who visited an emergency department due to CH was reported.
Time Frame: Week 4
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 100 | 104
Participants
  0 visits | 98 | 99
  1 visit | 1 | 2
  2 visits | 1 | 2
  3 visits | 0 | 1

27. Secondary Outcome: HCRU Score: Number of Hospital Admissions Due to Cluster Headache
Description: Number of participants who were admitted to a hospital due to CH was reported.
Time Frame: Week 4
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 100 | 104
Participants
  0 admissions | 97 | 102
  1 admission | 1 | 0
  2 admissions | 2 | 1
  3 admissions | 0 | 1

28. Secondary Outcome: HCRU Score: Number of Overnight Hospital Stays Due to Cluster Headache
Description: Number of participants who stayed overnight in a hospital due to CH was reported.
Time Frame: Week 4
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 100 | 104
Participants
  0 overnight hospital stays | 99 | 104
  5 overnight hospital stays | 1 | 0

29. Secondary Outcome: Change From Baseline in the Work Productivity Activity Impairment (WPAI) Questionnaire Subscores at Week 4
Description: The WPAI:GH2.0 is a patient self-rated clinical outcome assessment designed to provide a quantitative measure of the work productivity and activity impairment due to a health condition. The WPAI:GH2.0 assesses activities over the preceding 7 days and consists of 6 items: 1 item assesses employment (yes/no); 3 items assess the number of hours worked, the number of hours missed from work due to the participant's condition, or due to other reasons; and 2 visual numerical scales assess how much the participant's condition affects his/her productivity at work and his/her ability to complete normal daily activities. Each item (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) was calculated into an impairment percentage ranging from 0 to 100%, with higher numbers indicating greater impairment and less productivity (i.e. worse outcomes). Change from baseline for each item is shown here.
Time Frame: Baseline (Week 0), Week 4
Population: The APRS included all randomized participants. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure and "Number Analyzed" is the number of participants evaluable for each specified category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 95 | 95
score on a scale
  Absenteeism: number analyzed (Participants) | 65 | 66
  Absenteeism | -13.71 (3.95) | -4.37 (3.74)
  Presenteeism: number analyzed (Participants) | 57 | 56
  Presenteeism | -19.29 (4.81) | -11.03 (4.68)
  Work productivity loss: number analyzed (Participants) | 57 | 56
  Work productivity loss | -23.59 (5.34) | -13.68 (5.20)
  Activity impairment | -25.84 (3.70) | -15.82 (3.58)

ADVERSE EVENTS:
Time Frame: From date of first dose of IMP to 20 weeks after last dose (up to 24 weeks)
Description: The APTS included all randomized participants in the who received infusion with double-blind IMP.
Groups:
- Placebo-controlled Period: Eptinezumab: Participants received a single IV infusion of eptinezumab 400mg in 100 mL 0.9% saline solution.
- Placebo-controlled Period: Placebo: Participants received a single IV infusion of 0.9% saline solution as matching placebo for eptinezumab.
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo | Delayed Start Period: Eptinezumab to Placebo | Delayed Start Period: Placebo to Eptinezumab
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/117 | 0/108 | 0/107
Serious Adverse Events (participants affected / at risk) | 2/112 | 0/117 | 2/108 | 1/107
Other Adverse Events (participants affected / at risk) | 10/112 | 9/117 | 13/108 | 9/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-controlled Period: Eptinezumab (N=112) | Placebo-controlled Period: Placebo (N=117) | Delayed Start Period: Eptinezumab to Placebo (N=108) | Delayed Start Period: Placebo to Eptinezumab (N=107)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis enteroviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-controlled Period: Eptinezumab (N=112) | Placebo-controlled Period: Placebo (N=117) | Delayed Start Period: Eptinezumab to Placebo (N=108) | Delayed Start Period: Placebo to Eptinezumab (N=107)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (3) | 3 (4) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 7 (7) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04688775/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04688775/SAP_001.pdf